CLINICAL TRIAL: NCT06167629
Title: Monocentric Observational Study on the Diagnostic and Prognostic Role of 18F-PSMA PET (PET/CT and PET/MR) in Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: OMNIA_PSMA
Record Dates: First submitted 2023-11-24; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET 18F-PSMA — Subjects will be subjected to a PET examination according to international guidelines and where requested by the specialist. In particular, patients will be administered the radiopharmaceutical 18 F PSMA. Approximately two hours after administration, the patient is positioned on the PET/CT equipment table and image acquisition begins.

SUMMARY:
The general objective of this retrospective and prospective study is to evaluate the diagnostic and prognostic role of a quantitative analysis of PET images with 18F-PSMA in all stages of the disease in patients with prostate cancer. To this end, both imaging parameters commonly used in clinical practice and the contribution of radiomic features will be investigated. The latter are quantitative features extracted from biomedical images, and are believed to be able to provide information, otherwise impossible to investigate, useful for the characterization of various pathologies. This methodology is very promising, but also recent and therefore little studied and standardized. Our objective is also to investigate how to optimize it from a purely methodological point of view.

DETAILED DESCRIPTION:
In this study, all PET images with 18F-PSMA will be considered, but also the CT or MR images associated with them to allow better anatomical localization.

This study will allow us to investigate the diagnostic and prognostic role of l8F-PSMA PET, also evaluating its predictive value in terms of disease course, development of metastases and mortality. The retrospective part of this protocol is necessary for the acquisition of a sufficiently large amount of data to guarantee adequate statistical power for the study.

ELIGIBILITY:
Inclusion Criteria:

* adult male patients;
* patients with histopathological diagnosis of prostate cancer undergoing staging or restaging;
* patients with clinical indication for PET examination with 18 F-PSMA;

Exclusion Criteria:

* medical conditions that do not allow the acquisition of PET images;
* allergic reactions to iodinated contrast medium or creatinine levels >2mg/dL.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: The study will enroll adult patients with a histopathological diagnosis of prostate cancer undergoing PET examination with 18 F-PSMA where requested by the specialist due to clinical need at the U.O. of nuclear medicine of the San Raffaele Hospital.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2027-07-13 (Estimated); Study Completion 2027-07-13 (Estimated)

PRIMARY OUTCOMES:
PET with 18F-PSMA for diagnostic accuracy for staging of prostate cancer. | 5 years
  the role of a quantitative-semi-quantitative analysis for the characterization of prostatic pathology in different phases of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- IRC, Milan, Italy

IPD SHARING:
Plan to Share IPD: No